CLINICAL TRIAL: NCT05508750
Title: A Randomized, Controlled Trial Evaluating Growth and Safety in Infants Fed a New Infant Formula
Brief Title: Growth and Safety Clinical Trial on a New Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jovie USA, LLC (Industry)
Collaborators: IQVIA RDS Inc. (Industry); ObvioHealth (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IQV-JOV-001
Record Dates: First submitted 2022-08-18; First posted 2022-08-19 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Weight Gain
Keywords: infant; formula; in-home
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Intervention Model Description: A decentralized, randomized, controlled trial of healthy term breastfed and formula-fed infants for 16 weeks
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- New Infant Formula (Experimental): New infant formula for healthy term infants
  Interventions: Other: New Infant Formula
- Commercial Infant Formula (Active Comparator): Standard, commercially available infant formula for healthy term infants
  Interventions: Other: Commercial Infant Formula
- Human Milk (No Intervention): Breastfed infants serve as a reference group

INTERVENTIONS:
Other: New Infant Formula — New infant formula fed daily ad libitum
  Arms: New Infant Formula
Other: Commercial Infant Formula — Commercially available infant formula fed daily ad libitum
  Arms: Commercial Infant Formula

SUMMARY:
The aim of this study is to assess age-appropriate growth of healthy infants fed a new infant formula. In this randomized, controlled trial, healthy, term, formula-fed infants will be randomized to one of two infant formulas: a standard, commercially-available infant formula for term infants or the new infant formula for term infants for 16 weeks. A reference group of human milk-fed infants will also be enrolled. This study is designed in accordance with Good Clinical Practice guidelines and the requirements of the Code of Federal Regulations, 21CFR106.96. This study allows caregivers to participate completely from the comfort of their own home.

ELIGIBILITY:
Inclusion Criteria:

* Normal term infant (37-42 weeks gestation at birth)
* Infant <15 (+3) days of age at first study feeding, Birth constitutes day 0
* Infant birth weight of ≥2500 g (5.5 lbs.)
* Healthy Infant
* Caregiver who has previously decided to exclusively feed infant formula or exclusively breastfeed and is willing to continue with current feeding method throughout the study (breastfeeding or formula feeding)
* Caregiver willing to conform to protocol requirements (e.g. measuring, feeding, completion of food intake and tolerance diaries, and reporting of AEs)
* Caregiver willing and able to sign informed consent

Exclusion Criteria:

* Infant born in multiple birth (i.e., twins, triplets, etc.)
* Infant born with medical complications (e.g., neurological, cerebral palsy, etc.)
* Infant with family history (parents or siblings) of confirmed Milk or Soy allergies
* Infant with failure to thrive, fever, any GI tract abnormalities (e.g., short gut, gastroesophageal reflux, etc.), any congenital illness or malformation that may affect infant feeding or normal growth
* Caregiver intent to feed non-study formula or solid food during the study

Ages: 0 Days to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 420 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Weight gain from baseline to 16 weeks feeding | 16 weeks
  Weight gain g/day

SECONDARY OUTCOMES:
Length gain from baseline to 16 weeks feeding | 16 weeks
  Length gain
Head Circumference gain from baseline to 16 weeks feeding | 16 weeks
  Head Circumference gain
Volume of formula consumed during 3-consecutive day intervals | 16 weeks
  Volume of formula consumed

OTHER OUTCOMES:
Assessment of AEs | 16 weeks
  AEs reported during the study
Caregiver report of tolerance obtained during 3-consecutive day intervals | 16 weeks
  Caregiver report of fussiness, gassiness, and spitting up
Caregiver report of stool characteristics obtained during 3-consecutive day intervals | 16 weeks
  Caregiver report of stool consistency, color, and frequency
Stool collection for microbiome testing | 16 weeks
  Stool collection for microbiome testing at week 16 of feeding

CONTACTS AND LOCATIONS:
Overall Officials: Parth Shah, MD FAPCR, Principal Investigator — ObvioHealth; Dawn Ross, Director Clinical Project Management, Study Director — IQVIA RDS Inc.
Locations (1):
- ObvioHealth, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No